CLINICAL TRIAL: NCT00038506
Title: A Phase IV, Open-label, Multicenter Study of Treatment With TRIZIVIR (Abacavir 300mg/Lamivudine 150mg/Zidovudine 300mg) Twice Daily and Tenofovir 300mg Once-daily for 48 Weeks in HIV-infected Subjects Experiencing Early Virologic Failure (ZIAGEN Intensification Protocol)
Brief Title: Study Of Investigational Regimen Combining FDA Approved HIV Drugs In HIV Subjects Experiencing Early Virologic Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESS 30005
Record Dates: First submitted 2002-05-31; First posted 2002-06-03 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2010-10

CONDITIONS: HIV Infection
Keywords: HIV-1 TRIZIVIR Tenofovir
MeSH Terms: conditions — HIV Infections | interventions — abacavir, lamivudine, and zidovudine drug combination; Tenofovir

INTERVENTIONS:
Drug: abacavir/lamivudine/zidovudine
Drug: tenofovir
  Other Names: abacavir/lamivudine/zidovudine

SUMMARY:
This study is a 48-week study to evaluate the efficacy and safety of an investigational regimen combining FDA approved HIV drugs in antiretroviral-experienced subjects failing on their first highly active antiretroviral therapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Currently on an initial HAART (highly active antiretroviral therapy) regimen of 3TC/ZDV or 3TC/d4T and a PI (protease inhibitor) -boosted or unboosted- or NNRTI (non-nucleoside reverse transcriptase inhibitor).
* Plasma HIV - 1 RNA was <400 copies/ml on at least 2 documented occasions prior to viral rebound.
* Have a plasma HIV - 1 RNA value >400 copies/ml and <10,000 copies/ml on 2 documented successive occasions (including screen) separated by at least 2 weeks.
* A CD4+ lymphocyte count less than or equal to 100.

Exclusion Criteria:

* Have not taken Abacavir (ZIAGEN or TRIZIVIR) or tenofovir (VIREAD) previously.
* Have not had an AIDS defining illness within 30 days of screen.
* Pregnant or breast-feeding.
* Specified viral genotypes upon screening.
* And other inclusion or exclusion criteria to be evaluated by the physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-03; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
HIV viral load response at 48 weeks as measured by proportion of subjects with undetectable viral load. | 48 weeks

SECONDARY OUTCOMES:
Safety Viral load response at 24 weeks Change in T-cell count Resistance Health outcomes | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (25):
- United States (25):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Rafael, California
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Lake Worth, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Beach, Florida
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Maywood, Illinois
  - GSK Investigational Site, Lafayette, Indiana
  - GSK Investigational Site, Berkeley, Michigan
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Green Bay, Wisconsin